CLINICAL TRIAL: NCT01280721
Title: A Multicenter, Open-label Extension Study to Investigate the Long-term Safety and Efficacy of Tolvaptan in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) [Extension of Trial 156-04-251 in Japan]
Brief Title: A Study to Investigate the Long-term Safety and Efficacy of Tolvaptan in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) [Extension of Trial 156-04-251 in Japan]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-10-003; JapicCTI-101362 (Other: Japan Pharmaceutical Information Center)
Record Dates: First submitted 2010-12-06; First posted 2011-01-21 (Estimated); Results first posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2018-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease （ADPKD)
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tolvaptan (Experimental): Repeated oral administration twice daily (morning and evening) at one of three split dose-regimens 45mg/15mg, 60mg/30mg or 90mg/30mg.
  Interventions: Drug: tolvaptan

INTERVENTIONS:
Drug: tolvaptan — Repeated oral administration twice daily (morning and evening) at one of three split dose-regimens 45mg/15mg, 60mg/30mg or 90mg/30mg.

SUMMARY:
ADPKD patients who enrolled in Trial 156-04-251 will receive repeated oral administration of tolvaptan twice daily (morning and evening: 45mg/15mg, 60mg/30mg, or 90mg/30mg).

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in Trial 156-04-251 in Japan and for whom CRF collection has been completed.
* Patients who completed 3-year repeated administration and who completed the second follow-up visit or patients whose treatment with the trial drug was interupted due to pregnancy and who completed out the second follow-up visit in Trial 156-04-251.
* Patients in whom any adverse events occurring in Trial 156-04-251 were resolved orstabilized and require no further follow-up.

Exclusion Criteria:

* Patients with eGFR of less than 15 mL/min/1.73 m2
* Pregnant, breast-feeding, or possibly pregnant women or women who are planning to become pregnant
* Patients who received any investigational drug other than Tolvaptan within 30 days prior to commencement of administration of tolvaptan
* Any patients who, in the opinion of the principle investigator or subinvestigators, should not participate in the study

Ages: 23 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2010-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region

REFERENCES:
- [Derived] Muto S, Okada T, Yasuda M, Tsubouchi H, Nakajima K, Horie S. Long-term safety profile of tolvaptan in autosomal dominant polycystic kidney disease patients: TEMPO Extension Japan Trial. Drug Healthc Patient Saf. 2017 Oct 25;9:93-104. doi: 10.2147/DHPS.S142825. eCollection 2017. PMID 29123425

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolvaptan: Twice-daily repeated oral administration of tolvaptan at daily doses of 60 to 120 mg
Period: Overall Study
Arm/Group | Tolvaptan
Started | 135
Completed | 113
Not Completed | 22
Not completed — Adverse Event | 4
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 6
Not completed — eGFR under the withdrawal criteria | 7
Not completed — No tolerability for the lowest dose | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tolvaptan
Number analyzed (Participants) | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 58
Region of Enrollment [Number; unit: participants]
  Japan | 135

OUTCOME MEASURES:

1. Primary Outcome: Total Kidney Volume
Description: Measured values of total kidney volume (sum of the volume of the left and right kidneys) during trial period.
  Twice-daily repeated oral administration of tolvaptan at daily doses of 60 to 120 mg.
  Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, Month12, Month24, and Month36
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Baseline; Month 12; Month 24; Month 36: Measured values of total kidney volume (sum of the volume of the left and right kidneys) during trial period
Arm/Group | Baseline | Month 12 | Month 24 | Month 36
Number analyzed (Participants) | 135 | 123 | 120 | 27
mL | 1812.38 (859.21) | 1878.82 (950.60) | 1934.14 (926.79) | 2214.28 (842.87)

2. Primary Outcome: Renal Function Test (eGFR)
Description: Estimated glomerular filtration rate calculated by Japanese equation for eGFR during trial period.
  Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, Month12, Month24, and Month36
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Groups:
- Baseline; Month 12; Month 24; Month 36: Estimated glomerular filtration rate calculated by Japanese equation for eGFR during trial period
Arm/Group | Baseline | Month 12 | Month 24 | Month 36
Number analyzed (Participants) | 108 | 100 | 99 | 22
mL/min/1.73 m2 | 61.2 (21.7) | 56.3 (21.7) | 51.8 (20.1) | 43.5 (20.3)

3. Primary Outcome: Renal Function Test (Cys-C)
Description: Measured values of serum cystatin C concentration during trial period. Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, Month 12, Month 24, and Month 36
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Baselime; Month 12; Month 24; Month 36: Measured values of serum cystatin C concentration during trial period
Arm/Group | Baselime | Month 12 | Month 24 | Month 36
Number analyzed (Participants) | 108 | 100 | 99 | 22
mg/L | 1.016 (0.421) | 1.114 (0.477) | 1.129 (0.466) | 1.281 (0.461)

ADVERSE EVENTS:
Time Frame: Through study completion, 2 to 3 years for major patients
Arm/Group | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 0/135
Serious Adverse Events (participants affected / at risk) | 20/135
Other Adverse Events (participants affected / at risk) | 134/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=135)
Cardiac failure acute (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Umbilical hernias (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Renal cyst infection (Infections and infestations) | 4
Hepatic cyst infection (Infections and infestations) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Nasopharyngitis (Infections and infestations) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint dislocations (Injury, poisoning and procedural complications) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1
Renal pain (Renal and urinary disorders) | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 2
Renal cyst ruptured (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=135)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3
Palpitations (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Ventricular extrasystoles (Cardiac disorders) | 3
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 3
Vertigo (Ear and labyrinth disorders) | 3
Conjunctival haemorrhage (Eye disorders) | 5
Dry eye (Eye disorders) | 3
Glaucoma (Eye disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain lower (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 7
Dental caries (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 21
Enterocolitis (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 10
Chest pain (General disorders) | 5
Malaise (General disorders) | 5
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 8
Thirst (General disorders) | 104
Hepatic function abnormal (Hepatobiliary disorders) | 14
Hepatic steatosis (Hepatobiliary disorders) | 3
Seasonal allergy (Immune system disorders) | 5
Conjunctivitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 13
Hordeolum (Infections and infestations) | 4
Influenza (Infections and infestations) | 20
Nasopharyngitis (Infections and infestations) | 94
Pharyngitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Renal cyst infection (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 5
Arthropod sting (Injury, poisoning and procedural complications) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 5
Blood creatine phosphokinase increased (Investigations) | 6
Blood creatinine increased (Investigations) | 12
Blood pressure increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 3
Weight decreased (Investigations) | 8
Weight increased (Investigations) | 5
Hepatic enzyme increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 29
Dyslipidaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 30
Flank pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Dizziness (Nervous system disorders) | 10
Dizziness postural (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 26
Hypoaesthesia (Nervous system disorders) | 3
Intracranial aneurysm (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 8
Dysuria (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 6
Nocturia (Renal and urinary disorders) | 6
Pollakiuria (Renal and urinary disorders) | 77
Polyuria (Renal and urinary disorders) | 52
Renal cyst haemorrhage (Renal and urinary disorders) | 5
Renal impairment (Renal and urinary disorders) | 10
Dysmenorrhoea (Reproductive system and breast disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 6
Urticaria (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 20
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No